CLINICAL TRIAL: NCT02070549
Title: A Phase I Trial of Single Agent Trametinib (GSK1120212) in Advanced Cancer Patients With Hepatic Dysfunction
Brief Title: Trametinib in Treating Patients With Advanced Cancer With or Without Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00416; NCI-2014-00416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 9591; 9591/PJC-015; PJC-015; 9591 (Other: University Health Network Princess Margaret Cancer Center LAO); 9591 (Other: CTEP); N01CM00100 (NIH); U01CA132123 (NIH); U01CA062487 (NIH); U01CA062490 (NIH); UM1CA186644 (NIH); UM1CA186689 (NIH); UM1CA186690 (NIH); UM1CA186704 (NIH); UM1CA186709 (NIH); UM1CA186712 (NIH); UM1CA186717 (NIH); NCT02007382 (obsolete NCT alias)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Liver; Metastatic Malignant Solid Neoplasm; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase I trial studies the side effects and best dose of trametinib in treating patients with cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) with or without liver (hepatic) dysfunction. Trametinib may stop the growth of tumor cells by blocking proteins needed for cell growth. When these proteins are blocked, the growth of cancer cells may be stopped and the cancer cells will then die. Hepatic dysfunction is frequently found in patients with advanced cancer and usually prevents patients from receiving standard treatments or from participating in clinical trials. Patients may also need dose adjustments or absorb drugs differently. Trametinib may be a better treatment for patients with advanced cancers and hepatic dysfunction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide appropriate dosing recommendations for patients with varying degree of hepatic dysfunction receiving trametinib (mild, moderate and severe).

II. To establish the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of trametinib in advanced cancer patients with varying degrees of hepatic dysfunction.

III. To characterize the pharmacokinetic (PK) profile of trametinib in advanced cancer patients with varying degrees of hepatic dysfunction.

SECONDARY OBJECTIVES:

I. To document the non-DLTs associated with the administration of trametinib in patients with varying degrees of hepatic dysfunction.

II. To document any antitumor activity associated with trametinib treatment of patients enrolled on this study.

III. To explore and characterize predictive biomarkers for individual cancer patients utilizing genomic sequencing technologies.

OUTLINE: This is a dose-escalation study.

Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed solid malignancy that is metastatic or unresectable for which standard curative or palliative treatments do not exist or are no longer effective

  * Hepatocellular carcinoma (HCC) patients are not required to have histologically or cytologically confirmed malignancy, patients are considered eligible based on tumor markers and/or imaging assessment
  * Based on recent data that have shown limited trametinib benefit, patients with the following tumor types will be excluded from the normal and mild cohorts:

    * Pancreatic cancer patients
    * Colorectal cancer patients
    * BRAF V600E melanoma patients who have failed BRAF inhibitors

      * Note: Patients with pancreatic cancer, colorectal cancer, and BRAF V600E melanoma patients who have failed BRAF inhibitors are allowed to enroll in the moderate and severe cohorts provided the patients: 1) sign a separate consent form which outlines the extremely limited activity observed in prior studies, and 2) are consented to the study by a protocol-specified designee who is not their longitudinal oncologist
* All patients must have completed any prior chemotherapy, targeted therapy, radiotherapy (unless palliative doses which must be discussed with study principal investigator), surgery, anti-angiogenic therapy or interferon >= 28 days before study entry
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grade =< 1 (except alopecia) at the time of enrollment
* Absolute neutrophil count (ANC) >= 1.2 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 75 x 10^9/L
* Serum creatinine =< 1.5 mg/dL (=< 133 umol/L) OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Proteinuria =< +1 on dipstick or =< 1 gram/24 hours
* Prothrombin time (PT) =< 1.5 x institutional upper limit of normal (ULN)
* International normalized ratio (INR) =< 1.5 x institutional ULN
* Partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* No distinction should be made between liver dysfunction due to metastases and liver dysfunction due to other causes
* Patients with abnormal hepatic function will be eligible and will be grouped according to criteria summarized below:

  * Group A: Normal hepatic function

    * Bilirubin =< ULN
    * Aspartate aminotransferase (AST) =< ULN
  * Group B: Mild hepatic dysfunction

    * B1: bilirubin =< ULN and AST > ULN
    * B2: ULN < bilirubin =< 1.5 x ULN and any AST
  * Group C: Moderate hepatic dysfunction

    * 1.5 x ULN < bilirubin =< 3 x ULN and any AST
  * Group D: Severe hepatic dysfunction

    * 3 x ULN < bilirubin =< 10 x ULN and any AST; hepatic function tests should be repeated within 24 hours prior to starting initial therapy and may result in patients' group assignment being altered if different to registration test results
  * Patients with active hemolysis should be excluded. No distinction should be made between liver dysfunction due to metastases and liver dysfunction due to other causes. Hepatic function tests should be repeated within 24 hours prior to starting initial therapy and may result in patients' group assignment being altered if different to registration test results
* Trametinib can cause fetal harm when administered to a pregnant woman; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to registration and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of another malignancy

  * Exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 28 days prior to enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrollment
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib and during the study; patients previously treated with v-raf murine sarcoma (RAF) and/or mitogen-activated protein kinase (MEK) inhibitors are excluded from the study; multikinase antiangiogenic tyrosine kinase inhibitors such as regorafenib, sorafenib, sunitinib, etc. whose primary mechanism of action is not RAF inhibition, are allowed; if there are any questions, please contact study's principal investigator
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or excipients or to dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (Note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, PK, and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * LVEF < LLN
  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators
  * Known cardiac metastases
* Active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible)
* Patients with known human immunodeficiency virus (HIV) infection are eligible if not on antiviral agents and cluster of differentiation (CD)4 counts are adequate (>= 500)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Animal reproductive studies have not been conducted with trametinib; therefore, the study drug must not be administered to pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Any condition or medical problem in addition to the underlying malignancy and organ dysfunction which the investigator feels would pose unacceptable risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of trametinib | 28 days
  Dose escalation and determination of the maximum tolerated dose will be carried out separately for each cohort or stratum. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.
Dose-limiting toxicity | 28 days
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 beginning April 1, 2018). Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.
Pharmacokinetic profile of trametinib | Baseline and 0.5, 1, 2, 3, 4, 6, 10, and 24 hours on days 15 and 16 of cycle 1
  Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.

SECONDARY OUTCOMES:
Non-dose-limiting toxicities associated with the administration of trametinib | Up to 4 weeks post treatment
  Will document in patients with varying degrees of hepatic dysfunction.
Objective response to treatment | Up to 4 weeks post treatment
  Will be assessed using the Response Evaluation Criteria in Solid Tumors criteria 1.1. Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics.
Predictive biomarkers for individual cancer patients | Up to 4 weeks post treatment
  Will be assessed by utilizing genomic sequencing technologies. Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L Siu, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (11):
- United States (8):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas
- Canada (3):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Voon PJ, Chen EX, Chen HX, Lockhart AC, Sahebjam S, Kelly K, Vaishampayan UN, Subbiah V, Razak AR, Renouf DJ, Hotte SJ, Singh A, Bedard PL, Hansen AR, Ivy SP, Wang L, Stayner LA, Siu LL, Spreafico A. Phase I pharmacokinetic study of single agent trametinib in patients with advanced cancer and hepatic dysfunction. J Exp Clin Cancer Res. 2022 Feb 7;41(1):51. doi: 10.1186/s13046-021-02236-7. PMID 35130943